CLINICAL TRIAL: NCT01186861
Title: A Randomized, Double-Blind, Placebo-controlled Phase 2 Study of Maintenance OSI-906 Plus Erlotinib (Tarceva®), or Erlotinib Plus Placebo in Patients With Nonprogression Following Four Cycles of 1st-line Platinum-based Chemotherapy for Advanced NSCLC
Brief Title: Phase 2 Study of Maintenance OSI-906 Plus Erlotinib (Tarceva®), or Placebo Plus Erlotinib in Patients With Nonprogression Following 4 Cycles of Platinum-based Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OSI-906-205; 2010-020916-12 (EudraCT Number)
Record Dates: First submitted 2010-08-19; First posted 2010-08-23 (Estimated); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Non-Small Cell Lung Cancer (NSCLC) With Nonprogression Following 4 Cycles of Platinum-based Chemotherapy
Keywords: OSI-906; Erlotinib; Platinum-based chemotherapy; Placebo; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — 3-(8-amino-1-(2-phenylquinolin-7-yl)imidazo(1,5-a)pyrazin-3-yl)-1-methylcyclobutanol; Erlotinib Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: OSI-906 plus erlotinib (Experimental): OSI-906 150 mg twice daily (BID) starting on Day 1; erlotinib 150 mg once daily (QD) starting on Day 1
  Interventions: Drug: OSI-906; Drug: erlotinib
- Arm B: placebo plus erlotinib (Placebo Comparator): placebo BID starting on Day 1: erlotinib 150 mg QD starting on Day 1
  Interventions: Drug: erlotinib; Drug: placebo

INTERVENTIONS:
Drug: OSI-906 — Tablet administered with food and with up to 200 mL of water
  Arms: Arm A: OSI-906 plus erlotinib
Drug: erlotinib — Tablet administered at least 2 hours after food with up to 200 mL of water
  Other Names: OSI-774; Tarceva
Drug: placebo — Tablet administered at least 2 hours after food with up to 200 mL of water
  Arms: Arm B: placebo plus erlotinib

SUMMARY:
A multicenter, randomized, double-blind, placebo-controlled, phase 2 study with a 1:1 randomization scheme.

DETAILED DESCRIPTION:
Adult patients with advanced Non-small Cell Lung Cancer (NSCLC) and nonprogression after platinum-based chemotherapy will be randomized 1:1 to receive either OSI-906 plus erlotinib or placebo plus erlotinib.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed locally advanced or metastatic stage IIIB or IV NSCLC
* Have experienced Complete Response (CR), Partial Response (PR) or Stable Disease (SD) following completion of 4 cycles of first-line platinum-based chemotherapy and are not progressing at time of entry into study (prior completed first-line combination bevacizumab therapy is permitted; however, current use of maintenance bevacizumab is not permitted. A maximum interval of 28 days between the last day of the treatment cycle and randomization
* Patient has recovered from prior chemotherapy-related toxicity to ≤ grade 2
* EGFR mutation status must be confirmed for participation in the study. EGFR analysis can be performed either by central or local laboratory. If analysis is done locally, verifiable documentation confirming the EGFR mutation status must be submitted for review and approval by APGD prior to randomization. If no local result is available, formalin-fixed, paraffin-embedded archival tissue representative of the tumor or in the absence of archival tissue, a fresh tumor tissue sample of sufficient size to perform EGFR mutation analysis must be submitted centrally. Results of the central analysis must be available prior to randomization. Additionally, subjects should provide tissue blocks centrally for biomarker analysis whenever possible. Ideal tissue requirement: block with ≥5 mm2 tumor area sufficient to provide four 4-micron, and five 10-micron sections)
* Measurable disease (for those patients with PR or SD after first-line platinum-based chemotherapy) according to Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.1)
* Eastern Cooperative Oncology Group (ECOG) Performance Status(PS) 0 - 1
* Previous adjuvant or neo-adjuvant treatment is permitted
* Must be able to take oral medication
* Fasting glucose ≤ 150 mg/dL (8.3 mmol/L). Concurrent use of non-insulinotropic antihyperglycemic therapy is permitted if the dose has been stable for ≥ 4 weeks at the time of randomization
* Adequate hematopoietic, hepatic, and renal function defined as follows:

  * Neutrophil count ≥ 1.5 x 109/L
  * Platelet count ≥ 100 x 109/L
  * Bilirubin ≤ 1.5 x Upper Limit of Normal (ULN)
  * AST and ALT ≤ 2.5 x ULN, or ≤ 5 x ULN if patient has documented liver metastases
  * Serum creatinine ≤ 1.5 x ULN
* Potassium, magnesium and calcium within normal limits (supplementation and retesting is permitted)

Female patient must be either:

* Of non child bearing potential:

  * post-menopausal (defined as at least 1 year without any menses) prior to

Screening, or

* documented surgically sterile or status post hysterectomy (at least 1 month prior to Screening)

  * Or, if of childbearing potential:
* must have a negative urine pregnancy test at Screening, and
* must use two forms of birth control (one of which must be a barrier method) starting at Screening and throughout the study period and for 30 days after final study drug administration

  * Female patient must not be breastfeeding at Screening or during the study period and for 30 days after final study drug administration
  * Female patient must not donate ova starting at Screening and throughout the study period and for 30 days after final study drug administration
  * Male patient and their female spouse/partners who are of childbearing potential must be using highly effective contraception consisting of two forms of birth control (one of which must be a barrier method) starting at Screening and continue throughout the study period and for 30 days after final study drug administration
  * Male patient must not donate sperm starting at Screening and throughout the study period and for at least 30 days after final study drug administration
  * Prior radiation therapy is permitted provided patients have recovered from acute toxic effects of radiotherapy prior to randomization. A minimum of 28 days must have elapsed between the end of radiotherapy and randomization
  * Prior surgery is permitted provided that the surgery was performed 21 days prior to randomization and adequate wound healing has occurred prior to randomization
  * Patients must provide written (signed) informed consent to participate in the study and for use of tumor tissues

Exclusion Criteria:

* Prior exposure to agents directed at the Human Epidermal Receptor (HER) axis (eg, erlotinib, gefitinib, cetuximab, and trastuzumab)
* Malignancies other than NSCLC within past 3 years (exceptions if curatively treated: basal or squamous cell carcinoma of skin; locally advanced prostate cancer; ductal carcinoma in situ of breast; in situ cervical carcinoma; and superficial bladder cancer)
* Type 1 diabetes mellitus or Type 2 diabetes mellitus currently requiring insulinotropic or insulin therapy
* Prior insulin-like growth factor receptor (IGF-1R)
* Prior investigational agent within 21 days prior to randomization
* Concurrent use of maintenance bevacizumab
* History of poorly controlled gastrointestinal disorders that could affect the absorption of study drug (eg, Crohn's disease, ulcerative colitis, etc)
* History (within last 180 days) of significant cardiovascular disease unless the disease is well-controlled. Significant cardiac disease includes second/third degree heart block; clinically significant ischemic heart disease; superior vena cava (SVC) syndrome; poorly controlled hypertension; congestive heart failure of New York Heart Association (NYHA) Class II or worse (slight limitation of physical activity; comfortable at rest, but ordinary physical activity results in fatigue, palpitation, or dyspnea)
* History of arrhythmia (multifocal premature ventricular contractions [PVCs], bigeminy, trigeminy, ventricular tachycardia, or uncontrolled atrial fibrillation) that is symptomatic or requires treatment (≥ grade 3), left bundle branch block (LBBB), or asymptomatic sustained ventricular tachycardia are not allowed. Patients with atrial fibrillation controlled by medication are not excluded
* Mean QTcF interval > 450 msec based on independent central reviewer analysis of screening visit ECGs
* Use of drugs that have a known risk of causing Torsades de Pointes (TdP) are prohibited within 14 days prior to randomization
* Use of the potent CYP1A2 inhibitors ciprofloxacin and fluvoxamine. Other less potent CYP1A2 inhibitors/inducers are not excluded
* Use of potent CYP3A4 inhibitor such as ketoconazole, clarithromycin, atazanavir, indinavir, itraconazole, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, troleandomycin (TAO), or voriconazole
* Use of proton pump inhibitors such as omeprazole. Use of H2-receptor antagonists such as ranitidine are not excluded
* History of cerebrovascular accident (CVA) within 180 days prior to randomization or that resulted in ongoing neurologic instability
* Active infection, serious underlying medical condition (including any type of active seizure disorder within 12 months prior to randomization), or serious chronic illness that would impair the ability of the patient to receive study drug
* History of any psychiatric or neurologic condition that might impair the patient's ability to understand or to comply with the requirements of the study or to provide informed consent
* Pregnant or breast-feeding females
* Symptomatic brain metastases that are not stable, require steroids, or that have required radiation and/or other related treatment (e.g., anti-epileptic medication) within 21 days prior to randomization
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study drug
* Participated in any interventional clinical study or has been treated with any investigational drugs within 30 days or 5 half lives whichever is longer, prior to the initiation of Screening or during the course of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2011-03-04 (Actual); Primary Completion 2013-07-01 (Actual); Study Completion 2015-03-11 (Actual)

PRIMARY OUTCOMES:
The Progression Free Survival (PFS) of maintenance OSI-906 plus erlotinib, or placebo plus erlotinib in patients with nonprogression following four cycles of first-line platinum-based chemotherapy for advanced NSCLC in the overall population | 22 months
  PFS is defined as the time from randomization to disease progression based on RECIST v1.1 or death due to any cause whichever comes first

SECONDARY OUTCOMES:
Overall survival (OS) | 27 months
  The time from the date of randomization until the documented date of death
Disease control Rate (DCR) | 27 months
  The proportion of patients with a best overall response of continued Complete Response (CR), CR, Partial Response (PR), OR Stable Disease (SD) based on RECIST criteria
Best overall response rate (ORR) | 27 months
  The proportion of patients with a best overall response of CR or PR based on RECIST criteria
Response upgrade rate (RUR) | 27 months
  The proportion of patients with a response upgrade
Duration of response | 27 months
  The time from the date of the first documented response (CR/PR) to documented progression or death due to underlying cancer
Safety assessed through physical examination, vital signs, clinical laboratory tests, electrocardiograms (ECG) and Adverse Events | 27 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development
Locations (69):
- United States (7):
  - Site US10007, Jacksonville, Florida
  - Site US10001, Port Saint Lucie, Florida
  - Site US10002, Albany, Georgia
  - Site US10008, Chicago, Illinois
  - Site US10011, Scarborough, Maine
  - Site US10004, Greensboro, North Carolina
  - Site US10010, Winston-Salem, North Carolina
- Brazil (14):
  - Site BR55005, Barretos
  - Site BR55004, Brasília
  - Site BR55015, Cachoeiro de Itapemirim
  - Site BR55011, Florianópolis
  - Site BR55003, Fortaleza
  - Site BR55016, Goiânia
  - Site BR55006, Ijuí
  - Site BR55001, Itajaí
  - Site BR55008, Piracicaba
  - Site BR55013, Porto Alegre
  - Site BR55014, Porto Alegre
  - Site BR55012, Ribeirão Preto
  - Site BR55002, Rio de Janeiro
  - Site BR55007, São Paulo
- Canada (4):
  - Site CA11001, Oshawa
  - Site CA11004, Ottawa
  - Site CA11006, Toronto
  - Site CA11002, Toronto
- Germany (13):
  - Site DE49014, Berlin
  - Site DE49008, Cologne
  - Site DE49011, Dortmund
  - Site DE49003, Großhansdorf
  - Site DE49001, Heidelberg
  - Site DE49002, Hemer
  - Site DE49009, Homburg/Saar
  - Site DE49006, Immenhausen
  - Site DE49012, Karlsruhe
  - Site DE49015, Kassel
  - Site DE49010, Lübeck
  - Site DE49013, Mainz
  - Site DE49005, Minden
- Poland (4):
  - Site PL48002, Elblag
  - Site PL48005, Szczecin
  - Site PL48008, Torun
  - Site PL48006, Wroclaw
- Romania (7):
  - Site RO40005, Alba Iulia
  - Site RO40001, Baia Mare
  - Site RO40007, Brasov
  - Site RO40002, Cluj-Napoca
  - Site RO40003, Cluj-Napoca
  - Site RO40006, Craiova
  - Site RO40004, Hunedoara
- Russia (5):
  - Site RU70002, Chelaybinsk
  - Site RU70010, Kazan'
  - Site RU70007, Saint Petersburg
  - Site RU70009, Saint Petersburg
  - Site RU70011, Saint Petersburg
- South Korea (8):
  - Site KR82007, Busan
  - Site KR82006, Hwasun
  - Site KR82008, Incheon
  - Site KR82004, Seongnam-si
  - Site KR82003, Seoul
  - Site KR82005, Seoul
  - Site KR82002, Seoul
  - Site KR82001, Suwon
- United Kingdom (7):
  - Site GB44007, Bristol
  - Site GB44006, Dundee
  - Site GB44003, Leeds
  - Site GB44002, Leicester
  - Site GB44005, London
  - Site GB44001, Manchester
  - Site GB44004, Southampton

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency.

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=229